CLINICAL TRIAL: NCT04747561
Title: Clinical Application of 18F-PEG3-FPN PET Imaging in Diagnosis and Staging of Malignant Melanoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0016
Record Dates: First submitted 2021-02-07; First posted 2021-02-10 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-PEG3-FPN PET (Experimental): A positron probe for the targeted melanin
  Interventions: Drug: 18F-PEG3-FPN

INTERVENTIONS:
Drug: 18F-PEG3-FPN — For clinically suspected or confirmed melanoma patients and healthy volunteers, integrated PET/MR imaging was performed using targeted melanin-specific imaging agent 18F-PEG3-FPN. Meanwhile, the general imaging agent 18F-FDG was compared with MR multi-sequence and multi-parameters
  Other Names: 18F-FDG

SUMMARY:
This study is a diagnostic study. Patients and healthy volunteers were recruited from clinically suspected or confirmed melanoma patients to undergo 18F-PEG3-FPN PET/MR or PET/CT imaging to observe the response of the subjects after drug injection, and evaluate the efficacy of 18F-PEG3-FPN PET imaging in the diagnosis and staging of melanoma compared with 18F-FDG PET imaging. PET/CT imaging was performed in patients with contraindications to MR. The subjects underwent 18F-PEG3-FPN and 18F-FDG PET/MR or PET/CT imaging at an interval of two days, respectively. The general information, clinical data, blood routine, liver and kidney function indexes, 18F-PEG3-FPN and 18F-FDG PET/MR or PET/CT imaging results and other imaging data of the patients and volunteers were collected, and the histopathology of biopsy or surgical specimen was taken as the final diagnostic criteria. This study plans to set the sample size as 50 cases.

DETAILED DESCRIPTION:
This team always picolinamide structure based, successfully synthesized a positron nuclide targeting melanin probe - 18-5 - f FPN [18 f - 5 - fluoro - N - (2 - (diethyl amino) ethyl) pyridine formamide] for PET imaging, we found that combining FPN and melanin with high specificity and favorable pharmacokinetic characteristics, can be sensitive to detect the tiny metastases (lung, lymph node metastasis), which shows good potential of PET imaging for melanoma.The preparation method of 18F-5-FPN is simple and can be directly synthesized and purified by GE's synthesis module automatically.Then, we optimized the probe with triethylene glycol (PEG3), 18F-PEG3-FPN, to improve the labeling rate of the probe (44.68% >;6.98%, 18F-5-FPN), reduced its uptake in the liver, improved its drug distribution in vivo, and was successfully applied in the detection of liver metastasis.The integrated TOF PET/MR imaging equipment is the most advanced imaging equipment at present, which combines the advantages of PET and MR. With the high sensitivity of PET and the high soft tissue contrast of MR, it has obvious advantages over PET/CT in head, neck, abdomen and pelvic lesions.

At the same time, MR has no additional radiation and is more biosafety. With 18 f - PEG3 - FPN in clinical potential of melanoma imaging, 18 f - this project intends to apply PEG3 - FPN integrated PET/MR imaging diagnosis and staging of malignant melanoma tumors and clinical use of 18 f - FDG PET/CT imaging contrast, design of a prospective study, explore 18 f - PEG3 - FPN detection performance of melanoma, to make up for 18 f - FDG PET imaging diagnosis and staging of melanoma value.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 years or above), regardless of gender；
* Patients with clinically suspected or confirmed melanoma (supporting evidence including visual examination, MRI, CT, ultrasound, and histomathological examination, etc.) who agree to undergo histomathological examination (if not performed before imaging) and 18F-FDG PET imaging;Healthy volunteers;
* The patient or his legal representative can sign the informed consent.

Exclusion Criteria:

* Acute systemic diseases and electrolyte disturbances;
* Pregnant or lactating women;
* The patient or his legal representative is unable or unwilling to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 18F-PEG3-FPN PET/MR for diagnosis and staging in melanoma. | up to 2 years
  For subjects with suspected or diagnosed or treated melanoma who have completed 18F-FDG PET/CT imaging, diagnosis and staging results of 18F-PEG3-FPN PET/MR, PET/CT will be compared to 18F-FDG PET/CT imaging, pathology, clinical and follow-up result.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China